CLINICAL TRIAL: NCT01978821
Title: Open Label Study of Autologous Bone Marrow Mononuclear Cells in Cerebral Palsy
Brief Title: Stem Cell Therapy for Cerebral Palsy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-01
Record Dates: First submitted 2013-10-25; First posted 2013-11-08 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; autologous bone marrow mononuclear cells; stem cell therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell (Experimental): autologous bone marrow mononuclear cell transplantation
  Interventions: Procedure: Autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Procedure: Autologous bone marrow mononuclear cell transplantation

SUMMARY:
the purpose of this study was to study the effect of stem cell therapy on common symptoms of cerebral palsy patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of any type of Cerebral Palsy
* age above 12 months.

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* space occupying lesion in brain
* other acute medical conditions such as respiratory infection and pyrexia.

Ages: 17 Months to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in clinical symptoms of cerebral palsy after 6 months | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Li Y, Tu L, Chen D, Jiang R, Wang Y, Wang S. [Study on functional recovery of hypoxic-ischemic brain injury by Rg1-induced NSCs]. Zhongguo Zhong Yao Za Zhi. 2012 Feb;37(4):509-14. Chinese. PMID 22667154
- [Background] Sharma A, Sane H, Paranjape A, Gokulchandran N, Kulkarni P, Nagrajan A, Badhe P. Positron emission tomography-computer tomography scan used as a monitoring tool following cellular therapy in cerebral palsy and mental retardation-a case report. Case Rep Neurol Med. 2013;2013:141983. doi: 10.1155/2013/141983. Epub 2013 Feb 3. PMID 23431488
- [Background] Wang X, Cheng H, Hua R, Yang J, Dai G, Zhang Z, Wang R, Qin C, An Y. Effects of bone marrow mesenchymal stromal cells on gross motor function measure scores of children with cerebral palsy: a preliminary clinical study. Cytotherapy. 2013 Dec;15(12):1549-62. doi: 10.1016/j.jcyt.2013.06.001. Epub 2013 Oct 5. PMID 24100132
- [Background] Alvarez P, Carrillo E, Velez C, Hita-Contreras F, Martinez-Amat A, Rodriguez-Serrano F, Boulaiz H, Ortiz R, Melguizo C, Prados J, Aranega A. Regulatory systems in bone marrow for hematopoietic stem/progenitor cells mobilization and homing. Biomed Res Int. 2013;2013:312656. doi: 10.1155/2013/312656. Epub 2013 Jun 17. PMID 23844360